CLINICAL TRIAL: NCT03935815
Title: Quadratus Lumborum Nerve Blocks in Laparoscopic Myomectomy Patients
Brief Title: Quadratus Lumborum Nerve Blocks for Myomectomies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed prior to completion secondary to surgeon leaving UCLA
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Natale Naim, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-000825
Record Dates: First submitted 2019-02-26; First posted 2019-05-02 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Laparoscopic Myomectomy; Quadratus Lumborum Nerve Block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Standard of care pain management plus quadratus lumborum nerve block.
  Ropivicaine 0.25% 60 mL will be injected in the fascial plane between the quadratus lumborum muscle and transverses abdominus muscle.
  Interventions: Drug: Ropivacaine injection
- Control (Sham Comparator): Standard of care pain management plus a sham procedure.
  Interventions: Procedure: Sham treatment

INTERVENTIONS:
Drug: Ropivacaine injection — 30 mL of 0.25% ropivacaine will be administered on both the right and left sides with a 20 gauge, 4 inch ultrasound needle using a SonoSite ultrasound machine with a linear transducer probe. The tip of the ultrasound needle will be placed posterior to the quadratus lumborum muscle (QL2) made in the plane between the quadratus lumborum muscle and thoracolumbar fascia.
  Arms: Intervention
Procedure: Sham treatment — A sham procedure with a superficial 22 gauge needle stick will be performed without injectate.
  Arms: Control

SUMMARY:
This study would like to compare the use of the current standard of care in pain management for patients undergoing laparoscopic myomectomies to the addition of a quadratus lumborum nerve block plus the standard of care. Patients will be consented and the nerve blocks will be placed after the patients are placed under general anesthesia. Standard pain management will continue regardless of which arm of the study patients are in and measurements of pain scores, narcotic usage and abdominal numbness will be assessed in the post-operative period.

DETAILED DESCRIPTION:
This study aims to investigate benefits to the use of quadratus lumborum nerve blocks for laparoscopic myomectomies. Outcomes measured will be analgesic efficacy, incidence of post-operative events, patient satisfaction and narcotic usage.

Once a patient meets eligibility criteria and has consented to enter the study, randomization will be performed by the concealed envelope method. If chosen to be in the intervention group, a regional-trained anesthesiologist will perform the procedure, different from the intra-operative anesthesiologist. The control group will receive a superficial needle stick in the same location the quadratus lumborum block would have been otherwise placed.

Pre-operative protocol:

No premedications will be given while in the pre-operative waiting area. A member of the study group will randomly chose a concealed envelope indicating whether the patient will be in the control or intervention group.

Intraoperative protocol:

All patients will have standard ASA monitoring including: continuous electrocardiography, non-invasive blood pressure, percutaneous oxygen saturation, end-tidal carbon dioxide measurements, and heart rate.

Induction of general anesthesia and endotracheal intubation will be performed with propofol 1-2mg/kg and fentanyl 100 mcg. Dexamethasone 10mg IV will be administered for all patients for post-operative nausea risk reduction.

Maintenance of general anesthesia with be performed with sevoflurane 2-3% inhalation. Rocuronium 0.8-1 mg/kg intravenously will be administered for muscle relaxation.

After the patient is intubated and hemodynamically stable, the quadratus lumborum block procedure will be performed under ultrasound guidance by the regional trained anesthesiologist. First, a pillow or rolled blanket will be placed under the patient's hip for a semi-lateral position. 30 mL of 0.25% ropivacaine will be administered on both the right and left sides with a 20 gauge, 4 inch ultrasound needle using a SonoSite ultrasound machine with a linear transducer probe. The tip of the ultrasound needle will be placed posterior to the quadratus lumborum muscle (QL2) made in the plane between the quadratus lumborum muscle and thoracolumbar fascia.

After performing the block, intra-operative fentanyl administration will be at the discretion of the intraoperative anesthesiologist. On surgical closure, acetaminophen 1000 mg IV and ketorolac 15mg IV will be administered. No long acting opioids (eg hydromorphone, morphine) will be given intra-operatively. Ondansetron 4mg IV will be administered for post-operative nausea risk reduction. Sugammadex 2 mg/kg will be administered for reversal of neuromuscular blockade. Extubation will be performed by the intra-operative anesthesiologist.

Post-operative Protocol:

Patients will be asked their pain scores at rest and with movement at the designated time intervals: Arrival to PACU (t=0), 1 hr, 2hr, 3hr, and at PACU discharge. Severity of pain will be on a 10-point Numeric Rating Scale (NRS 0 = no pain, NRS 10 = worst imaginable pain).

A worksheet will be given to the patient at discharge and the patient will fill out her pain score 6 hours, 24 hours, and 48 hours after surgery. Nursing staff will ask and record pain scores while in the PACU in the electronic medical system. A study member will make phone calls home after PACU discharge to collect data from the patient.

While in the PACU, all patients will be ordered for intravenous fentanyl 25 mcg for mild pain, fentanyl 50 mcg for moderate pain, fentanyl 100 mcg for severe pain.

Patients will be ordered for oxycodone PO 5mg for mild pain, oxycodone PO 10mg for moderate pain, oxycodone PO 15 mg for severe pain while in the recovery room.

All patients will be discharged home with the same prescription of oxycodone 5mg, one pill every 4 hours as needed. All patients will be instructed to take acetaminophen 650mg every 6 hours by mouth for the first 24 hours (6 doses, total 2,600 mg for 24 hours) as needed.

It is currently not the standard of care to place these regional anesthesia nerve blocks, but we do think they offer great value and are hoping to produce results which will change what the standard of care entails.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1-2,
* Female,
* greater than or equal to 18 years of age,
* undergoing laparoscopic myomectomy surgery

Exclusion Criteria:

* History of chronic pain requiring preoperative opioids,
* congenital coagulopathy,
* anatomic abnormalities,
* localized soft tissue infection,
* use of anticoagulants,
* unable to comprehend pain scoring system,
* severely obese (BMI > 35)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Morphine equivalents (MOE) consumption | Up to 24 hours after surgery
  The patient's cumulative intake of morphine over 24 hours.

SECONDARY OUTCOMES:
Pain Score | Up to 48 hours after surgery
  Rate of pain on a scale of 0-10 (0 is no pain and 10 is the worst pain possible)

CONTACTS AND LOCATIONS:
Locations (1):
- Ronald Reagan UCLA Medical Center, Department of Anesthesiology, Los Angeles, California, United States

REFERENCES:
- [Result] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Result] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Result] Carvalho R, Segura E, Loureiro MD, Assuncao JP. [Quadratus lumborum block in chronic pain after abdominal hernia repair: case report]. Rev Bras Anestesiol. 2017 Jan-Feb;67(1):107-109. doi: 10.1016/j.bjan.2014.08.001. Epub 2014 Dec 6. Portuguese. PMID 25487690
- [Result] Visoiu M, Yakovleva N. Continuous postoperative analgesia via quadratus lumborum block - an alternative to transversus abdominis plane block. Paediatr Anaesth. 2013 Oct;23(10):959-61. doi: 10.1111/pan.12240. Epub 2013 Aug 9. PMID 23927552
- [Result] Chakraborty A, Goswami J, Patro V. Ultrasound-guided continuous quadratus lumborum block for postoperative analgesia in a pediatric patient. A A Case Rep. 2015 Feb 1;4(3):34-6. doi: 10.1213/XAA.0000000000000090. PMID 25642956